CLINICAL TRIAL: NCT00952302
Title: Physiology Study Investigating the Effects of Supplementation and Depletion of Iron on Hypoxia-related Pulmonary Hypertension
Brief Title: Study of the Effects of Iron Levels on the Lungs at High Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Ms Heather House, Head of Clinical Trials and Research Governance, University of Oxford
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Oxford-Peru-2008
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Pulmonary Hypertension; Mountain Sickness
Keywords: Hypoxia; Iron; Hypoxia-Inducible Factor 1; Chronic mountain sickness
MeSH Terms: conditions — Hypertension, Pulmonary; Altitude Sickness; Hypoxia | interventions — Ferric Oxide, Saccharated; Saline Solution; Phlebotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CMS - placebo first (Placebo Comparator): Patients with chronic mountain sickness (CMS) who are venesected and studied for several weeks. In the final crossover period of the study, patients receive a placebo (saline) infusion first followed by iron infusion.
  Interventions: Procedure: Venesection; Drug: Iron sucrose; Drug: Normal saline
- CMS - iron (Experimental): Patients with chronic mountain sickness (CMS) who are venesected and studied for several weeks. In the final crossover period of the study, patients receive an iron infusion first followed by placebo (saline) infusion.
  Interventions: Procedure: Venesection; Drug: Iron sucrose; Drug: Normal saline
- SLR - placebo (Placebo Comparator): Sea level residents (SLR) taken to high altitude for one week, and receiving placebo (saline) infusion on Day 3 at high altitude.
  Interventions: Drug: Normal saline
- SLR - iron (Experimental): Sea level residents (SLR) taken to high altitude for one week, and receiving iron infusion on Day 3 at high altitude.
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: Iron sucrose — Single intravenous infusion of iron 200 mg
  Other Names: Venofer
  Arms: SLR - iron
Drug: Normal saline — Single intravenous infusion of normal 0.9% saline 100 mls (as placebo)
  Arms: SLR - placebo
Procedure: Venesection — Isolvolaemic venesection of total 2 litres of blood - 500 mls each day for 4 days, replaced with normal saline.
  Arms: CMS - iron; CMS - placebo first
Drug: Iron sucrose — Two intravenous infusions, each of 200 mg of iron, separated by one day.
  Other Names: Venofer
  Arms: CMS - iron; CMS - placebo first
Drug: Normal saline — Two intravenous infusions of normal 0.9% saline 100 mls (as placebo), separated by one day.
  Arms: CMS - iron; CMS - placebo first

SUMMARY:
The study hypothesis is that body iron levels are important in determining the increase in lung blood pressure that occurs in response to low oxygen levels. The purpose of this study is to determine whether this is true at high altitude, where oxygen levels are low.

DETAILED DESCRIPTION:
Pulmonary hypertensive disorders frequently complicate hypoxic lung disease and worsen patient survival. Hypoxia-induced pulmonary hypertension is also a major cause of morbidity at high altitude. Hypoxia causes pulmonary hypertension through hypoxic pulmonary vasoconstriction and vascular remodelling. These processes are thought to be regulated at least in part by the hypoxia-inducible factor (HIF) family of transcription factors, which coordinate intracellular responses to hypoxia throughout the body.

HIF is regulated through a cellular degradation process that requires iron as an obligate cofactor. In cultured cells HIF degradation is inhibited by reduction in iron (by chelation with desferrioxamine) and potentiated by iron supplementation. In humans, we have recently shown that, in laboratory experiments lasting 8 hours, acute iron supplementation blunts the pulmonary vascular response to hypoxia, while acute iron chelation with desferrioxamine enhances the response.

This suggests that iron may also affect the pulmonary artery pressure response to hypoxia over longer time periods. The purpose of this study is to investigate this link between iron and the pulmonary artery pressure response to hypoxia, through a study conducted at high altitude allowing concurrent exposure of larger numbers of participants to environmental hypoxia. We wish to explore the extent and the time-course of the effect of iron on pulmonary artery pressure. Cerro de Pascu (4,340 m) in Peru provides the unique ability to make rapid transitions from sea level to high altitude (6-8 hours by road), together with the requisite research facilities. Also, one part of this study involves recruitment of patients with chronic mountain sickness, of whom there are many living in Cerro de Pasco.

ELIGIBILITY:
SLR ARM

Inclusion Criteria:

* sea level natives of lowland ancestry
* generally in good health
* detectable tricuspid regurgitation on echocardiography

Exclusion Criteria:

* any significant medical problem
* known susceptibility to high altitude pulmonary or cerebral oedema
* taking medications or iron supplements

CMS ARM

Inclusion Criteria:

* diagnosis of chronic mountain sickness
* no recent venesection therapy (within 1 year)
* detectable tricuspid regurgitation on echocardiography

Exclusion Criteria:

* any other significant medical problem

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary artery systolic pressure | One week (SLR arm) and one month (CMS arm)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Robbins, BMBCh DPhil, Principal Investigator — University of Oxford
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Peru

REFERENCES:
- [Derived] Smith TG, Talbot NP, Privat C, Rivera-Ch M, Nickol AH, Ratcliffe PJ, Dorrington KL, Leon-Velarde F, Robbins PA. Effects of iron supplementation and depletion on hypoxic pulmonary hypertension: two randomized controlled trials. JAMA. 2009 Oct 7;302(13):1444-50. doi: 10.1001/jama.2009.1404. PMID 19809026